CLINICAL TRIAL: NCT00502736
Title: An Open Label Study to Assess the Effect of Intravenous Loading Doses of Bondronat on Bone Pain in Patients With Breast Cancer and Skeletal Metastases
Brief Title: A Study of Loading Doses of Intravenous Bondronat (Ibandronate) in Patients With Breast Cancer and Malignant Bone Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20684
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Bone Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bondronat]

INTERVENTIONS:
Drug: ibandronate [Bondronat] — 6mg iv on days 1-3

SUMMARY:
This single arm study will assess the efficacy and safety of loading doses of intravenous Bondronat in patients with breast cancer and malignant bone disease experiencing moderate to severe bone pain. Patients will receive an intravenous infusion of 6mg Bondronat on days 1, 2 and 3. The anticipated time on study treatment is 3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* breast cancer;
* bone metastases;
* moderate to severe pain;
* adequate renal function.

Exclusion Criteria:

* bisphosphonate treatment within 3 weeks of study enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain and analgesic consumption | Days 1, 7 and 14

SECONDARY OUTCOMES:
AEs and laboratory parameters | Days 1, 4 and 7
Serum creatinine | Days 1, 4 and 7
Karnofsky index | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Shhiye, Ankara